CLINICAL TRIAL: NCT04000620
Title: The Role of CNN Architecture-based Transfer Learning of Medical Imaging in Lung Cancer Diagnosis and Staging
Brief Title: Imaging-based Deep Learning for Lung Cancer Diagnosis and Staging
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Yang Jin, Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: AFDSFA
Record Dates: First submitted 2019-06-24; First posted 2019-06-27 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cancer cell involvement predicted by deep learning: the participants with lesions of lung, lymph node or other sites predicted as positive for cancer cell involvement by imaging based deep learning.
  Interventions: Procedure: surgery; Procedure: punture
- no cancer cell involvement predicted by deep learning: the participants with lesions of lung, lymph node or other sites predicted as negative for cancer cell involvement by imaging based deep learning.
  Interventions: Procedure: surgery; Procedure: punture

INTERVENTIONS:
Procedure: surgery — treatment intent surgery
Procedure: punture — diagnostic punture

SUMMARY:
Lung cancer diagnosis and staging are two fundamental and critical issue in clinical lung cancer management and therapeutic decision-making. Invasive procedures for pathologic analysis are gold standard for diagnosis and staging, however, invasive procedures related-complications are inevitable. Noninvasive medical imaging is a powerful tool, however there is almost no room for improvement just according to the experience of radiologist and clinician. The researchers will investigate the role of computer based deep learning of medical imaging in the diagnosis of lesion of lung, lymph node and other sites suspected with metastasis.

DETAILED DESCRIPTION:
Radiologist

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of lung cancer
* PET/CT or CT examination before any cancer-specific treatment

Exclusion Criteria:

* A history of other malignancies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung cancer patients with PET/CT or CT examination before any cancer-specific treatment
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
pathologic result revealed cancer cell involvement in lesion | 1 month after the pathologic test

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided